CLINICAL TRIAL: NCT02414126
Title: Evaluation of Breathing, Sleep and the Effects of Continuous Positive Airway Pressure During Wakefulness in Children With Heart Failure
Acronym: IC-E-PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Philips Healthcare (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014 A1907-40
Record Dates: First submitted 2015-02-24; First posted 2015-04-10 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart failure; child; work of breathing; cardiac function; sleep; polysomnography; CPAP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Children with dilated cardiomyopathy with an ejection fraction (Active Comparator)
  Interventions: Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness; Device: CPAP
- Children with univentricular congenital heart disease (Active Comparator)
  Interventions: Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness; Device: CPAP
- Children with left valvulopathy (Active Comparator)
  Interventions: Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness; Device: CPAP

INTERVENTIONS:
Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness — Comparison of three periods of 3 hours
  1. st period: Spontaneous breathing for 10 minutes
  2. nd period: CPAP for 10 minutes
  3. rd period: Spontaneous breathing for 10 minutes to check the return to baseline.
  After each period, the following parameters will be recorded during 5 minutes:
  * oesogastric pressures
  * air flow
  * gas exchange
  * right and left cardiac function
  Patients > 6 years old will assess their dyspnea on a visual analogue scale
  Arms: Children with dilated cardiomyopathy with an ejection fraction
Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness — Comparison of three periods of 3 hours
  1. st period: Spontaneous breathing for 10 minutes
  2. nd period: CPAP for 10 minutes
  3. rd period: Spontaneous breathing for 10 minutes to check the return to baseline.
  After each period, the following parameters will be recorded during 5 minutes:
  * oesogastric pressures
  * air flow
  * gas exchange
  * right and left cardiac function
  Patients > 6 years old will assess their dyspnea on a visual analogue scale
  Arms: Children with univentricular congenital heart disease
Other: Effect of CPAP on respiratory work and cardiac function indices during wakefulness — Comparison of three periods of 3 hours
  1. st period: Spontaneous breathing for 10 minutes
  2. nd period: CPAP for 10 minutes
  3. rd period: Spontaneous breathing for 10 minutes to check the return to baseline.
  After each period, the following parameters will be recorded during 5 minutes:
  * oesogastric pressures
  * air flow
  * gas exchange
  * right and left cardiac function
  Patients > 6 years old will assess their dyspnea on a visual analogue scale
  Arms: Children with left valvulopathy
Device: CPAP

SUMMARY:
Adult patients with heart failure (HF) have an increased work of breathing and are at increased risk for obstructive and/or central apnea during sleep. Noninvasive continuous positive airway pressure (CPAP) has proved its efficacy in decreasing the work of breathing and improving sleep-disordered breathing in these patients.

The aim of the study is to analyze the work of breathing and objective and subjective sleep quality in children with HF and to evaluate the ability of noninvasive CPAP to decrease the work of breathing and improve cardiac output during wakefulness.

DETAILED DESCRIPTION:
The study starts with the measurement during wakefulness of

* the breathing pattern and work of breathing
* and cardiac function during 5 min after 10 min of stable and calm spontaneous breathing (SB) Then the same measurement are made during 5 min after 10 min of stable and calm breathing during non-invasive CPAP Then a third measurement is made of
* the breathing pattern and work of breathing
* and cardiac function during 5 min after 10 min a stable and calm SB

Polysomnography is then performed during the following night during SB in order to assess objective sleep quality.

Subjective sleep quality is assessed on the following morning in children > 6 years of age by validated sleep questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A child with HF and having:
* Dilated cardiomyopathy with an ejection fraction <45%
* Univentricular congenital heart disease
* Left ventricular valvulopathy
* Age 8 months to 17 years
* Signed informed consent by the owner (s) of parental authority and investigator
* Patient affiliated to a social security scheme or entitled (excluding MEAs)
* Comparison of results depending on the status T21 / T21 not.

Exclusion Criteria:

* HF with use of inotropic drugs during the last 30 days.
* Contra indication to CPAP or inability to maintain the airway or adequately remove phlegm, risk of aspiration of gastric contents, acute sinusitis or diagnosis of otitis media, epistaxis, hypotension.
* Associated pathology may be responsible alone an obstructive apnea (ENT or maxillofacial malformation pathology, abnormalities of the upper airway, obesity with BMI z-score> 2), a central apnea syndrome (Chiari malformation), or alveolar hypoventilation (neuromuscular disease, cystic fibrosis or bronchopulmonary dysplasia).

Ages: 8 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
oesophageal pressure during spontaneous breathing and during continuous positive airway pressure | up to 5 days
trans-diaphragmatic pressure during spontaneous breathing and during continuous positive airway pressure | up to 5 days

SECONDARY OUTCOMES:
Ultrasound cardiac function indices during spontaneous breathing and during continuous positive airway pressure | up to 5 days
Polysomnography during spontaneous breathing | up to 5 days
sleep questionnaire | up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Necker - Enfants Malades Hospital (Assistance Publique des Hopitaux de Paris), Paris, France

REFERENCES:
- [Background] Amaddeo A, Khraiche D, Khirani S, Meot M, Jais JP, Bonnet D, Fauroux B. Continuous positive airway pressure improves work of breathing in pediatric chronic heart failure. Sleep Med. 2021 Jul;83:99-105. doi: 10.1016/j.sleep.2021.04.003. Epub 2021 Apr 19. PMID 33991896